CLINICAL TRIAL: NCT03847558
Title: Assessment of Sexual Maturation in β-Thalassemia Major Patients Receiving Iron Chelation Therapy in Assiut University Hospital
Brief Title: Sexual Maturation in β-Thalassemia Major Patients in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ayman ekram, Principal Investigator, Assiut University
Other Study IDs: Assiut Univ Children Hospitals
Record Dates: First submitted 2018-12-04; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: β-Thalassemia Major Patients Receiving Chelation Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sexual maturation in patient receiving iron chelation: assess of sexual maturation by clinical examination and hormonal studies (FSH.LH,Testosterone)
  Interventions: Diagnostic Test: FSH((Follicle Stimulating Hormone) and LH (Luteinizing Hormone) hormone for females and Testosterone hormone for males

INTERVENTIONS:
Diagnostic Test: FSH((Follicle Stimulating Hormone) and LH (Luteinizing Hormone) hormone for females and Testosterone hormone for males — assess of sexual maturation by clinical examination and hormonal studies (FSH.LH,Testosterone)

SUMMARY:
cross sectional study to asses sexual maturation in β-Thalassemia Major patients receiving Iron Chelation Therapy in assuit University Hospital and maintenance of 2ry sexual characters and reproduction

DETAILED DESCRIPTION:
Thalassemia refers to a group of inherited diseases characterized by decreased or absent synthesis of normal globin chains . The direct consequence is an imbalance of the alpha and beta globin chain synthesis that results in anemia from ineffective erythropoiesis and hemolysis.

The term thalassemia major refers to the severe form that is often associated with life-long transfusion dependent anemia.

Hypogonadism is the most frequently reported endocrine complication, affecting 70-80% of thalassemia major patients. Hypogonadism is likely to be caused by iron deposits in the gonads, pituitary gland or both.

Hypogonadotropic hypogonadism resulting from iron deposition in the pituitary gonadotrope is more commonly found than gonadal iron deposition in ovaries or testes occurs.

Iron deposition in the anterior pituitary gland can be demonstrated beginning in the first decade of life, but clinical manifestations are usually not evident until the onset of puberty. At the earlier stage, only a diminished gonadotropin reserve with intact gonadotropin pulse was observed .

The direct effect of iron, in particular that of NTBI(non-transferrin-bound iron) on the ovaries and testes is currently unknown. The ovarian reserve is preserved in the majority of female thalassemia patients, even in women with amenorrhea. In males, histological examination of testicular tissues from autopsies demonstrated testicular interstitial fibrosis with small, heavily pigmented, undifferentiated seminiferous tubules and an absence of Leydig cells .

There are three main clinical presentations of the HPG(hypothalamic pituitary gonadal axis)axis derangement in thalassemia major, including delayed puberty, arrested puberty and hypogonadism. Delayed puberty is defined as the absence of any pubertal signs by 14 years in boys and 13 years in girls . Arrested puberty is defined as the absence of further pubertal progression for more than 1 year after puberty has started.

Chelation therapy with desferoxamine before the age of puberty has helped patients to attain normal sexual maturation in some studies but not in others. In a study of 40 patients with transfusion-dependent thalassemia major, 90% of 19 patients who began treatment with desferoxamine before the age of 10 had normal sexual development compared with only 38% of those treated after the age of 10. In contrast, another study reported no difference in the frequency of pubertal maturation when iron chelation therapy was started at the age of 10 or earlier. Serum ferritin levels were still higher than normal in previous studies.

After a period of 5-7 years, 50% of hypogonadal males achieved normal testosterone levels and 32% of amenorrheic women became pregnant, either spontaneously or using in vitro fertilization . With modern medications, iron-induced hypogonadism may be reversible with intensive iron chelation regimens.

ELIGIBILITY:
Inclusion Criteria:

* β-thalassemic Patients aged 10 years and older
* β-thalassemic patients receiving regular blood transfusions
* All patients are on chelation therapy

Exclusion Criteria:

* β-thalassemic patients with major system complications as cardiac ,renal or hepatic.
* Patients not receiving chelation therapy
* Patients with other hemolytic anemia

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: β-thalassemic Patients aged 10 years and older patients receiving regular blood transfusions in Assiut Univ Hospitals and have chelation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
sexual maturation in patients receiving regular chelation will be compared to patients not receiving chelation helps us to improve quality of life for these patients and have normal sexual life | 1 year
  The present study will be carried out on previously diagnosed transfusion dependent thalassemia patients under chelation therapy in Assiut University children hospital.
  1. patients will be selected and examined clinically to asses thier sexual maturation by measuring presence of secondary sexual characters.
  2. hormonal assesment for patients including FSH,LH,Serum Testosterone.
calculate body mass index (kg/m^2) | 1 year
  assesment of hieght in meters,weight in kilograms.

IPD SHARING:
Plan to Share IPD: Undecided
i hope i can publish my study to help other researchers to get accurate assesment and improve reproduction of these patients